CLINICAL TRIAL: NCT06840847
Title: Sexual Coercion in Breast Cancer Patients Treated With Luteinizing Hormone-Releasing Hormone Agonists (LHRHa )
Acronym: LHRHa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canan Kas (Other)
Responsible Party: Sponsor-Investigator, Canan Kas, PhD, MSc, RN, Assistant Professor, Kastamonu University
Organization: Kastamonu University (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-KAEK-148; Kastamonu Universty 2023/148 (Other Grant/Funding Number: Kastamonu Universty)
Record Dates: First submitted 2025-02-01; First posted 2025-02-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: breast cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LHRHa (Active Comparator): In this study, included 40 patients on LHRHa. The instrument assessed partner sexual coercion in three domains: resource manipulation/sexual coercion, commitment manipulation, and threat of separation.
  Interventions: Behavioral: Sexual Coercion
- Tamoxifen (Nolvadex) (Active Comparator): In this study included 39 patients on tamoxifen. The instrument assessed partner sexual coercion in three domains: resource manipulation/sexual coercion, commitment manipulation, and threat of separation.
  Interventions: Behavioral: Sexual Coercion

INTERVENTIONS:
Behavioral: Sexual Coercion — This study aimed to investigate whether patients receiving LHRHa treatment experienced sexual coercion at a higher rate than those using tamoxifen. 40 patients using LHRHa and 39 patients using tamoxifen were included in the study.

SUMMARY:
The use of luteinizing hormone-releasing hormone agonists(LHRHa) to suppress ovarian function is a common strategy for treating premenopausal, hormone receptor-positive breast cancer. However, this approach can lead to more severe and prolonged menopausal symptoms, which can further impact intimate relationships and sexual function. Sexual coercion, encompassing both overt and subtle forms of pressure, is a significant global public health concern that threatens individual well-being.

DETAILED DESCRIPTION:
Objective: The use of luteinizing hormone-releasing hormone agonists(LHRHa) to suppress ovarian function is a common strategy for treating premenopausal, hormone receptor-positive breast cancer. However, this approach can lead to more severe and prolonged menopausal symptoms, which can further impact intimate relationships and sexual function. Sexual coercion, encompassing both overt and subtle forms of pressure, is a significant global public health concern that threatens individual well-being.

Methods: This study is a randomized controlled study. In this study, the validated Turkish version of the Sexual Coercion in Intimate Relationship Scale was utilized to investigate whether patients receiving LHRHa therapy experienced higher rates of sexual sexual coercion compared to those taking tamoxifen. The study included 40 patients using LHRHa and 39 patients using tamoxifen. The instrument assessed partner sexual coercion across three subdomains: resource manipulation/sexual coercion, commitment manipulation, and defection threat.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years of age
* willingness to participate in this study
* having received treatment for breast cancer
* having a history of breast cancer surgery
* having an active relationship with a spouse or partner.

Exclusion Criteria:

* having any neuropsychiatric disorder
* having any mental illness
* having a history of gynecological surgery
* currently receiving active chemotherapy or less than 3 months since completing chemotherapy
* receiving treatment for metastatic disease
* The use of selective serotonin reuptake inhibitors

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
LHRHa | for 10 months
  It was examined whether patients receiving LHRHa treatment were exposed to sexual pressure.
Tamoxifen | for 10 months
  It was examined whether patients receiving tamoxifen treatment were exposed to sexual pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Kastamonu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No